CLINICAL TRIAL: NCT04853446
Title: Oral Dexamethasone as an Adjunct to a Brachial Plexus Block in Patients Undergoing Orthopaedic Surgery of the Forearm and Hand. A Randomised, Blinded, Placebo-controlled, Parallel, Triple-arm Clinical Trial.
Brief Title: Oral Dexamethasone as an Adjunct to a Brachial Plexus Block in Patients Undergoing Orthopaedic Surgery of the Forearm and Hand
Acronym: ADJUNCT1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADJUNCT1
Record Dates: First submitted 2021-04-19; First posted 2021-04-21 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia, Local
Keywords: Peripheral nerve block; Dexamethasone; Adjunct; Regional anesthesia
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial medication was produced by Glostrup Pharmacy. The trial medication is produced as identically appearing opaque capsules containing either dexamethasone or placebo. The trial medication is stored in sequentially numbered containers that will be allocated to each participant as they enter the trial. All involved in the trial will be masked to treatment allocation until the final statistical analysis has been agreed upon by the steering committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Encapsulated glucosemonohydrate will be used as placebo. Two capsules containing placebo will be administered in the placebo arm.
  Interventions: Drug: Placebo
- Dexamethasone 12 mg (Experimental): Dexamethasone tablets of 4 mg encapsulated in pairs of three. One capsule containing 12 mg dexamethasone and one capsule containing placebo will be administered in the 12mg dexamethasone arm for a total dose of 12 mg of dexamethasone.
  Interventions: Drug: Dexamethasone 12 mg
- Dexamethasone 24 mg (Experimental): Dexamethasone tablets of 4 mg encapsulated in pairs of three. Two capsules containing 12 mg dexamethasone will be administered in the 25mg dexamethasone arm for a total dose of 24 mg of dexamethasone.
  Interventions: Drug: Dexamethasone 24 mg

INTERVENTIONS:
Drug: Dexamethasone 12 mg — Two identically appearing, opaque capsules will be administered: one capsule containing 12 mg of dexamethasone and one capsule containing placebo.
  Arms: Dexamethasone 12 mg
Drug: Placebo — Two identically appearing, opaque capsules will be administered: two capsules containing placebo.
  Arms: Placebo
Drug: Dexamethasone 24 mg — Two identically appearing, opaque capsules will be administered: two capsules each containing 12mg dexamethasone.
  Arms: Dexamethasone 24 mg

SUMMARY:
The investigators will assess the beneficial and harmful effects of oral dexamethasone (12 mg or 24 mg) versus placebo in patients undergoing orthopaedic surgery of their hand or forearm with a lateral infraclavicular brachial plexus block as the means of providing anaesthesia and analgesia.

DETAILED DESCRIPTION:
This is a randomised, blinded, placebo-controlled, multicentre, parallel, 3-arm clinical trial assessing the effects of adjunct oral dexamethasone (12mg or 24mg) versus placebo on time to first pain (i.e. block duration) in patients undergoing surgery of the forearm or hand. At the initiation of the trial, no other trials had examined the effects of oral dexamethasone as an adjunct to peripheral nerve blocks.

The investigators will randomise participants to either oral dexamethasone 12mg, oral dexamethasone 24mg, or placebo. Participants will be allocated according to a computer-generated random allocation sequence with random permuted blocks and stratification by site. Glostrup Pharmacy produced the trial medication and sequentially numbered the drug containers, thereby concealing the allocation.

All involved will be blinded for the entire duration of the trial (participant, carers, investigators, people delivering the intervention, observers/outcome assessors, statisticians). Blinding will not be broken until agreement has been reached within the steering committee regarding the statistical analysis. The trial medication is produced as identically appearing opaque capsules containing either dexamethasone or placebo. The trial medication is contained within identically appearing, sequentially labelled containers.

The investigators expect little to no attrition bias since the intervention is simple with a short follow-up. The investigators expect some missing data for duration of the motor block, as most participants will have the affected limb immobilized post-surgery, thereby making assessment of return of motor function difficult.

The investigators pre-defined the statistical analysis plan prior to unblinded data becoming available. The analysis plan can be found on: https://doi.org/10.6084/m9.figshare.22491214.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral osseous surgery of the hand or forearm.
* Anaesthesia with an infraclavicular brachial plexus block
* Age of 18 or above
* American Society of Anaesthesiologists Physical Status Score of 1 to 3
* Body Mass Index of 18 to 40, but a minimum weight of 50 kg.
* For fertile women, negative urine humane choriongonadotropine test and use of safe anti-conception
* Ability to understand the trial protocol, risks and benefits, and provide signed informed consent

Exclusion Criteria:

* Inability to read and understand Danish
* Uncooperativeness (as judged by investigators)
* Participation in another trial involving medication
* Allergy to study medication
* Daily use of opioids above 30 mg/day morphine (or equivalents)
* Daily use of corticosteroids of more than 5 mg prednisolone equivalents within the past one month
* Neurological or musculoskeletal disease making block performance impossible (as judged by investigators)
* Dysregulated diabetes (as judged by investigators)
* Dysregulated anti-coagulants (as judged by investigators)
* History of drug or alcohol abuse
* Glaucoma
* Contraindications for paracetamol or opioids
* Other concomitant conditions needing surgery
* Other concomitant traumatic injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Time to first pain (measured in minutes) | 48 hours
  Time to first pain will be recorded by the patient and measured as the time to first perceived pain in minutes in the surgical area. The patient will be asked to record the time and date of their first perceived pain in their trial log. This date and time will be compared to the date and time of the block performance as recorded in the electronic Case Report Form. In the event of the patient not experiencing any pain, the time to first pain will be set to 48 hours.

SECONDARY OUTCOMES:
Duration of the motor block (measured in minutes) | 48 hours
  Duration of the motor block will be recorded by the patient and measured in minutes as the time from removal of the needle to the first movement of their bicep muscle on the operative site, and not the first movement of their distal extremity. The patient will record the date and time of their time to first bicep movement on the operative side in their trial log. This date and time will be compared to the date and time of the block performance as registered in the electronic Case Report Form. In the event of the patient not regaining movement of the bicep, the duration of the motor block will be set to 48 hours.
Quality of sleep (Numerical Rating Scale) postoperative night 1 | 24 hours
  Sleep will be measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to the worst possible sleep and '10' points correspond to the best possible sleep. This outcome measure will be recorded by the patients in their trial log after the first postoperative night.
Quality of sleep (Numerical Rating Scale) postoperative night 2 | 48 hours
  Sleep will be measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to the worst possible sleep and '10' points correspond to the best possible sleep. This outcome measure will be recorded by the patients in their trial log after the second postoperative night.
Proportion of participants with one or more serious adverse events. | 30 days
  Serious adverse events as defined by the ICH-GCP will be collected and reported as the proportion of participants with one or more serious adverse events. Furthermore, the individual serious adverse events will also be reported.
Proportion of participants with one or more adverse events not considered to be serious | 48 hours
  We will record any adverse events not considered to be serious. We will report the proportion of participants with one or more adverse events not considered to be serious and all individual adverse events not considered to be serious.

OTHER OUTCOMES:
Cumulative oxycodone consumption (measured in milligrams) at 24 hours | 24 hours
  Cumulative oxycodone consumption will be recorded in the electronic medical files of the patients during hospitalisation and in their trial log at 24 hours and 48 hours by the patient after discharge. The patient will be instructed to record whenever they ingest escape oxycodone, as well as record the total amount of ingested escape oxycodone at 48 hours postoperatively. The patient will be instructed to not count in any usual opioid consumption, but only the escape oxycodone provided by the investigators.
Cumulative oxycodone consumption (measured in milligrams) at 48 hours | 48 hours
  Cumulative oxycodone consumption will be recorded in the electronic medical files of the patients during hospitalisation and in their trial log at 24 hours and 48 hours by the patient after discharge. The patient will be instructed to record whenever they ingest escape oxycodone, as well as record the total amount of ingested escape oxycodone at 48 hours postoperatively. The patient will be instructed to not count in any usual opioid consumption, but only the escape oxycodone provided by the investigators.
Pain (measured on the Numerical Rating Scale) at 24 hours postoperatively | 24 hours
  Pain will be recorded during rest and measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain. The patients will record their perceived pain at 24 hours postoperatively in their trial log.
Average pain (measured on the Numerical Rating Scale) from 0 to 24 hours postoperatively | 24 hours
  Participants will judge their average pain from 0 to 24 hours postoperatively as measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain.
Worst pain (measured on the Numerical Rating Scale) from 0 to 24 hours postoperatively | 24 hours
  Participants will judge their worst pain from 0 to 24 hours postoperatively as measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain.
Pain (measured on the Numerical Rating Scale) at 48 hours postoperatively | 48 hours
  Pain will be recorded during rest and measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain. The patients will record their perceived pain at 48 hours postoperatively in their trial log.
Average pain (measured on the Numerical Rating Scale) from 24 to 48 hours postoperatively | 48 hours
  Participants will judge their average pain from 24 to 48 hours postoperatively as measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain.
Worst pain (measured on the Numerical Rating Scale) from 24 to 48 hours postoperatively | 48 hours
  Participants will judge their worst pain from 24 to 48 hours postoperatively as measured on the Numerical Rating Scale from '0' to '10' points where '0' points correspond to no pain and '10' points correspond to the worst possible pain.
Patient satisfaction (added after initiation of the trial, will only be available for a subset of the patients) | 48 hours
  Patients will be inquired about their satisfaction with a peripheral nerve block related to:
  1. Pain during block performance (Numerical Rating Scale (NRS) from 0 to 10).
  2. Discomfort associated with having a blocked extremity (NRS from 0 to 10, 0 no discomfort & 10 worst discomfort).
  3. Pain immediately after block cessation (NRS from '0' to '10').
  4. Overall satisfaction with block (NRS from 0 to 10, 0 worst & 10 best).
  5. If the participant would accept a block in the future (yes/no)
  6. If the participant would recommend a block to others (yes/no).
  7. If the block duration was too long, too short, or adequate.
  8. Satisfaction with content of information regarding block (NRS 0 to 10, 0 worst & 10 best)
  9. Satisfaction with the amount of information regarding block (NRS 0 to 10, 0 worst & 10 best)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Maagaard, MD, Principal Investigator — Department of Anaesthesiology, Zealand University Hospital, Køge, Denmark
Locations (3):
- Denmark (3):
  - Department of Anaesthesiology, Køge, Zealand Region of Denmark
  - Department of Anaesthesiology, Slagelse, Zealand Region of Denmark
  - Department of Anaesthesiology, Bispebjerg Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data in anonymised form will be shared upon reasonable request to the primary investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When the trial has been completed, data analysed, and trials results published.
Access Criteria: Individual patient data in anonymised form will be shared upon reasonable request to the primary investigator.